CLINICAL TRIAL: NCT07212127
Title: Analgesic Effect of Transcutaneous Electrical Nerve Stimulation Based on Wrist-Ankle Acupuncture Theory Combined With Tramadol Hydrochloride During Oocyte Retrieval Surgery
Brief Title: Analgesic Effect of TENS-WAA Combined With Tramadol Hydrochloride During Oocyte Retrieval Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University (Other)
Responsible Party: Principal Investigator, Xiaonan Huang, researcher, First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHEC2025-347
Record Dates: First submitted 2025-09-19; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Oocyte Retrieval for IVF; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Before the trial begins, envelopes containing sequentially numbered cards from 1 to 60 will be prepared to determine participant allocation. The coordinator will open the envelopes in the order of participant enrollment. Throughout the trial, researchers are not allowed to alter the enrollment sequence. Participants will be informed in advance that they may experience electrical stimulation sensations, and communication between participants will be prohibited during the entire trial process. The statistician responsible for data analysis will remain blinded to the group allocation of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation Group (Experimental): According to the WAA theory, the selected Lower Zone 1 (LZ1) and Lower Zone 2 (LZ2) are defined as follows: LZ1 is located between the medial Achilles tendon and the medial malleolus, while LZ2 is positioned at the central inner edge of the ankle joint, near the posterior border of the tibia. Two electrode pads will be placed on each LZ1 and LZ2 of both legs, totaling eight electrode pads. The TENS-WAA device will be set to a frequency of 2 Hz, a pulse width of 500 μs, and a continuous waveform.The experimental group will receive transcutaneous electrical nerve stimulation based on wrist-ankle acupuncture theory 30 minutes prior to oocyte retrieval surgery, with current intensity adjusted to the maximum tolerable level. Tramadol hydrochloride 100mg will be administered intramuscularly 20 minutes before surgery.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory（TENS-WAA)
- Sham electrical stimulation group (Placebo Comparator): Participants in the control group will have the electrodes placed in the same positions as those in the stimulation group,with identical electrical stimulation frequency and pulse width settings.However,the control group received sham stimulation at the lowest intensity under identical conditions.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory（TENS-WAA)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory（TENS-WAA) — Based on the theory of wrist and ankle needles, transcutaneous electrical nerve stimulation is a kind of analgesic treatment device that combines wrist and ankle needles with transcutaneous electrical nerve stimulation, and can be worn on the human wrist and ankle. Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture Theory uses low-frequency electronic pulses to stimulate the entry point of the wrist-ankle needle, which has the advantages of easy to wear, concentration of the treatment site, safety of the treatment, and no needles.

SUMMARY:
This study is a single-centre randomised controlled trial. It aimed to evaluate the efficacy and safety of transcutaneous electrical nerve stimulation based on wrist-ankle acupuncture theory(TENS-WAA) combined with tramadol hydrochloride for analgesia during transvaginal ultrasound-guided oocyte retrieval, by comparing the analgesic effects and the prevention of postoperative nausea and vomiting between the TENS-WAA combined with tramadol hydrochloride group (experimental group) and the sham TENS-WAA combined with tramadol hydrochloride group (control group). Participants were randomly assigned to the experimental or control group. The experimental group received percutaneous electrical nerve stimulation based on wrist-ankle acupuncture theory 30 minutes prior to the procedure, at a frequency of 2Hz with current intensity adjusted to the maximum tolerable level.Tramadol hydrochloride 100mg was administered intramuscularly 20 minutes before surgery. The control group received sham stimulation at the lowest intensity under identical conditions. The primary outcome measure was the Visual Analogue Scale (VAS). Secondary outcome measures included skin conductance response, postoperative nausea scale, and vomiting scale.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 21 and 42 years.
* Patients diagnosed with infertility requiring oocyte retrieval for in vitro fertilisation-embryo transfer.
* Body Mass Index (BMI) 18.5 ≤ BMI ≤ 29.9 kg/m².
* Regular menstrual cycles with ultrasound monitoring demonstrating dominant follicle development and ovulation during the natural cycle; good ovarian reserve: follicle-stimulating hormone (FSH) < 10 IU/L, antral follicle count (AFC) > 6, anti-Müllerian hormone (AMH) > 1.5 ng/ml.
* Undergoing ovarian stimulation therapy using follicle-stimulating hormone (FSH) or gonadotropin protocols.
* Electing tramadol hydrochloride injection for analgesia during oocyte retrieval.
* Voluntary participation with signed written informed consent.

Exclusion Criteria:

* History of other chronic pain conditions, or prolonged use of opioid medications, history of anaesthetic drug addiction, or chronic alcohol abuse.
* Severe pelvic adhesions.
* Presence of pacemakers or other implanted medical electronic devices.
* Concurrent use of high-frequency surgical equipment, artificial heart-lung machines, medical shortwave therapy, or microwave therapy devices.
* Presence of scarring or skin lesions at electrode application sites.
* Severe anxiety, depression, or other psychiatric conditions impairing accurate description of sensations, or any other disorders potentially affecting pain perception.
* Conditions contraindicating or affecting oocyte retrieval, such as coagulation disorders, acute pelvic inflammation, vaginitis, trichomoniasis, endometriomas, ovarian cysts.
* Individuals with laparoscopically and/or ultrasonographically confirmed endometriosis.
* Patients with ovarian hyporesponsiveness following conventional ovarian stimulation medication.

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-08 (Estimated); Primary Completion 2026-11-08 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain VAS score | Within 3 minutes following oocyte retrieval
  VAS is used to assess pain. It is widely used in clinical practice in China. The basic method is to use a 10-cm long floating ruler with 10 scale marks on one side, with 0 and 10 marks at the two ends. 0 means no pain, and 10 means the most severe pain that is unbearable.

SECONDARY OUTCOMES:
Galvanic Skin Response | during procedure
  Galvanic Skin Response (GSR) is a bio-signal detection technique that reflects autonomic nervous system activity by measuring changes in skin conductance. Its core principle lies in the following: when an individual experiences emotional fluctuations, sympathetic nervous system excitation stimulates increased secretion from eccrine sweat glands. The electrolytes in sweat significantly alter the conductive properties of the skin surface, and these transient changes in conductance form the characteristic spikes of the GSR signal.
Nausea Rating Scale | 30 minutes after oocyte retrieval
  The Nausea Assessment Scale is divided into four scores: 0 points (None) indicates no nausea sensation; 1 point (Mild) indicates a feeling of wanting to vomit but without muscle contractions; 2 points (Moderate) indicates spasmodic contractions of the diaphragm and chest/abdominal muscles but without expulsion of gastric contents; 3 points (Severe) indicates frequent muscle contractions with expulsion of gastric contents.
Vomiting Rating Scale | 30 minutes after oocyte retrieval
  The Vomiting Assessment Scale is divided into four scores: 0 points (None) indicates no vomiting; 1 point (Mild) indicates vomiting 1-2 times; 2 points (Moderate) indicates vomiting 3-4 times; 3 points (Severe) indicates vomiting more than 5 times with expulsion of large amounts of gastric contents.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code